CLINICAL TRIAL: NCT05787600
Title: The Anti-inflammatory and Anti-plaque Efficacies of Mouth Rinse Containing Hyaluronic Acid and Hydrogen Peroxide in the Management of Dental Biofilm-induced Gingivitis: a 14 Days Randomized Clinical Trial
Brief Title: Anti-inflammatory and Anti-plaque Efficacies of Mouth Rinse Containing Hyaluronic Acid and Hydrogen Peroxide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ahmed Hashim Alyasari, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 748622
Record Dates: First submitted 2023-03-03; First posted 2023-03-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Plaque Induced Gingivitis; Mouth Diseases; Bleeding Gum; Periodontal Diseases
Keywords: Gingivitis; Plaque; Hyaluronic acid; hydrogen peroxide
MeSH Terms: conditions — Mouth Diseases; Gingival Hemorrhage; Periodontal Diseases; Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: 54 subjects with plaque induced gingivitis, caused by accumulation of plaque, will be selected and enrolled in this study. Subsequently, subjects will be equally divided and randomly allocated for three groups, each group received a similar number of subjects (n=18) with a 1:1:1 allocation.
Who Masked: Participant, Investigator
Masking Description: The products will be packaged in such a way that they are not recognizable neither by the operator, nor by the patient. Each package will be assigned a number that in turn will refer to the type of the product. The association between the number and type of the product will be collected by another operator according to the association carried out by a dedicated software. The operator who will deliver the product will be informed about the type only at the end of the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perhyal rinse (Experimental): Participants will be given the test interventions,Perhyal rinse, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing.
  Interventions: Drug: Perhyal rinse
- Chlorhexidine 0.12% (Active Comparator): Participants will be given the positive-control, Chlorhexidine 0.12%, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing.
  Interventions: Drug: Chlorhexidine mouthwash
- Placebo Product (Placebo Comparator): Participants will be given the nonactive control, distilled water, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perhyal rinse — Filming mouthwash formulation, enriched with Hydrogen Peroxide and Hyaluronic Acid Subjects will then be given the test intervention, Perhyal rinse, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE). No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 14 days.
  Other Names: BMG0703
  Arms: Perhyal rinse
Drug: Chlorhexidine mouthwash — Subjects will then be given Chlorhexidine 0.12%mouthwash, as an active comparator, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE). No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 14 days.
  Other Names: Chlorhexidine 0.12%
  Arms: Chlorhexidine 0.12%
Drug: Placebo — Subjects will be given the nonactive control, distilled water, and will be asked to rinse with 10 ml of undiluted mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE). No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 14 days.
  Other Names: Placebo product
  Arms: Placebo Product

SUMMARY:
The goal of this clinical trial is to test efficiency of using mouth rinse containing (H2O2 and HA) over a period of two weeks to control on gingival inflammation and plaque accumulation through measuring the clinical periodontal parameters (Gingival Index (GI), Bleeding on probing (BOP) and modified Quigley-Hein Plaque Index (mQHPI ) in comparison with Chlorhexidine (CHX) and placebo mouth rinses in patients with biofilm induced gingivitis.

Objectives:

* Evaluate the clinical efficiency of using mouth rinse containing (H2O2 and HA) over a period of 14 days to control on gingival inflammation and plaque accumulation through measuring the clinical periodontal parameters (Gingival Index, Bleeding on probing and modified Quigley-Hein Plaque Index in comparison with Chlorhexidine and placebo mouth rinses in patients with biofilm induced gingivitis.
* Measuring levels of salivary cytokines, Interleukin 1 beta (IL-1B) and Interleukin 6 (IL-6) at baseline visit before using mouth rinse and after 14 days of using the mouth rinse containing H2O2 and HA compared to chlorhexidine and placebo mouth rinses.
* Evaluate subjects' perception of a mouth rinse (H2O2 and HA), CHX and placebo mouth rinses after 14 days from using three mouth rinse

DETAILED DESCRIPTION:
54 subjects will be enrolled, who show with generalized gingivitis (having >30% bleeding sites with no PPD >3 mm, intact periodontium and no loss of periodontal attachment), caused by accumulation of plaque.

A double-blind, randomized parallel 3-arms clinical trial include using the following mouth rinses, 0.12% CHX (KIN Gingival, KIN, Barcelona, Spain) as positive-control , distilled water (placebo, nonactive control) with food additives (to blind the subjects and examiner) and Perhyal rinse (BMG Pharma, Milan, Italy ) containing has H2O2 (1,80%) and HA (0,10%) with the remaining part being water (97,3%) and inert additives as active ingredients, will be used as test interventions. The mouthwashes will be contained in identical opaque bottles that were randomly given sequential letters codes (A, B and C ) by a another subject who will not involved in the clinical investigation. This ensured the double blindness of both the participant and examiner during the clinical trial. Decoding will performed after the end of the study.

Randomization will be performed by the examiner for enrollment patient in 3 groups. Each group will be assigned a letter (A, B or C) corresponding to the intervention used. Random numbers were generated and used to re-sort the order of the groups and participants (n=54), who will distributing into designated groups, each group received a similar number of subjects (n=18) with a 1:1:1 allocation, by using a Microsoft Excel random table (Microsoft Office 2016, Microsoft Corporation, USA). Then, coded bottles with the interventions will be delivered to the participants together with instructions for use. The participants will be asked to rinse with 10 ml of undiluted.

mouthwash for 60 s twice per day (30 min after tooth brushing) and will be instructed to refrain from eating and drinking for 30 min after rinsing. Discontinuation of the mouthwash will be advised in cases of any allergic reaction. All participants will be received a toothbrush with medium-hardness bristles and a toothpaste (COLGATE®, Colgate-Palmolive, NY, USA). No modifications to the participants' tooth brushing technique will be permitted.

In baseline visit at the beginning,

Saliva collection for IL-1β and IL-6 measurement then clinical periodontal parameters examination starting with gingival index (Loe and Silness in 1963) designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed on the basis of color, consistency and bleeding on probing. A periodontal probe will be runned along the gingival margin. The gingiva surrounding the tooth is assessed at four sites: mesio-facial papilla, facial marginal gingiva, disto-facial papilla and lingual marginal gingiva.

Followed by dryness and wait then measurement of BOP for the six surfaces of all teeth except wisdom teeth through gently inserting the periodontal probe to the depth of the gingival sulcus then removed coronally and waited for 30 s to observe the presence of bleeding (0=no bleeding, 1=presence of bleeding)

Then finally followed by the Modified Quigley Hein Plaque Index with Fluorescein disclosing tablets. In the (mQHPI) the data had been recorded from labial/buccal and lingual/palatal surfaces of each disclosed tooth except wisdom teeth and any teeth had filling surface.

The distance from the gingival margin to the edge of the disclosed area measured to the nearest 0.5 mm using a calibrated periodontal probe and the scores registered according to record form of mQHPI for each participant. The mean of mQHPI for each participant had been calculated by collecting the scores over the total number of surfaces examined.

First visit after 14 days, from the baseline visit.

Saliva collection and clinical periodontal parameters scoring (GI, BOP ,mQHP) will be performed again as described at baseline visit. The mouthwash bottles will be retrieved, and the remaining volume will be determining to further evaluate the compliance with mouth rinsing.

(the total volume/bottle for two weeks will be 280 ml).

For the purpose of self-assessment, a visual analog scale (VAS)- score based questionnaire was filled out by each participant at the end of the trial to evaluate the intervention. The questionnaire and method of data interpretation were adopted and modified from a previous study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years-old.
* participants who were apparently systemically healthy.
* Presence of ≥ 20 teeth.
* Patients with generalized gingivitis (having >30% bleeding sites with no PPD >3 mm, intact periodontium and no loss of periodontal attachment .
* Patients without presence of supra- or subgingival calculus

Exclusion Criteria:

* Patients who refuse to write an informed consent form.
* Extensive untreated dental caries and diseases of hard and soft palate.
* Those having periodontitis.
* Ongoing orthodontic treatment.
* History of antibiotics intake within the past 3 months.
* Pregnant or intended to and lactating mother.
* Smoker or alcoholism
* Using mouthwash within past one month.
* Those with a recent tooth extraction.
* Those having a history of hypersensitivity to any product used in the present study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Gingival index | 0, 14 days
  Subjects will undergo the measurement of gingival index according to Loe & Silness, designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed on the basis of color, consistency and bleeding on probing. The gingiva surrounding the tooth is assessed at four sites: mesio-facial papilla, facial marginal gingiva, disto-facial papilla and lingual marginal gingiva. Data will be collected based on four possible clinical conditions:
  0=Normal gingiva1=Mild Inflammation-Slight change in color, Slight odema. No bleeding on probing2=Moderate inflammation-redness,odema and glazing. Bleeding on probing 3=Sever inflammation-marked redness and edema.Ulceration.Tendency to spontaneous bleeding.

SECONDARY OUTCOMES:
Mean amount plaque between different comparators. | 14 days
  Mean amount plaque between different comparators as anti-plaque agent after rinsing with different comparators using means of modified quigely hein plaque index[ Turesky ,1970]
Assessment of the interventions by the participants through answering specially designed | 14 days
  All subjects received a questionnaire using a visual analog scale(VAS) designed to evaluate their attitudes with regard to the product used. Subjects marked a point on a 10-cm-long uncalibrated line with the negative extreme response (0) at the left end and the positive extreme response (10) at the right end.
Mean relative changes in Interleukin 1 beta and Interleukin 6 levels in salivary Fluid. | 14 days
  Mean relative changes in Interleukin 1 beta and Interleukin 6 levels in salivary fluid after rinsing with different comparators from baseline at 14 days.
Changes in BOP score | 14 days
  For recording BOP score, the periodontal probe was inserted with gentle force into the sulcus/pocket until minimal resistance was felt. The probing force presumably was ranging between 20 to 25g. The examination started from the distal surface of the right upper 7 moving mesially to measure all the existing teeth. For each tooth, 6 surfaces were examined; the surface that displayed bleeding on probing was scored 1 and the surface with no bleeding was scored 0

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed alyasari, B.D.S, Principal Investigator — University of Baghdad
Locations (1):
- University of Baghdad\ College of Dentistry, Baghdad, Bab Al-Moadham, Iraq